CLINICAL TRIAL: NCT01976650
Title: Safety and Efficacy of Dexamethasone (OZURDEX®) Intravitreal Implant in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 206207-029
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: Patients who receive dexamethasone 700 ㎍ (OZURDEX®) intravitreal implant treatment for Branch Retinal Vein Occlusion, Central Retinal Vein Occlusion, or non-infectious uveitis affecting the posterior segment of the eye as per local standard of care in clinical practice.
  Interventions: Drug: dexamethasone 700 ㎍ intravitreal implant

INTERVENTIONS:
Drug: dexamethasone 700 ㎍ intravitreal implant — dexamethasone 700 ㎍ (OZURDEX®) intravitreal implant treatment for Branch Retinal Vein Occlusion, Central Retinal Vein Occlusion, or non-infectious uveitis affecting the posterior segment of the eye as per local standard of care in clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This study is a Post-Market Surveillance study in Korea to evaluate the safety and efficacy of dexamethasone 700 ㎍ (OZURDEX®) intravitreal implant used to treat Branch Retinal Vein Occlusion, Central Retinal Vein Occlusion, or non-infectious uveitis affecting the posterior segment of the eye in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Branch Retinal Vein Occlusion, Central Retinal Vein Occlusion, or non-infectious uveitis affecting the posterior segment of the eye treated with (OZURDEX®) in clinical practice.

Exclusion Criteria:

* Patients with eye infections
* Patients with glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Branch Retinal Vein Occlusion, Central Retinal Vein Occlusion, or non-infectious uveitis affecting the posterior segment of the eye treated with (OZURDEX®) in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Kim MS, Choi J, Lee HD, Woo SJ; Korea Ozurdex Post-Marketing Surveillance Study Group. Dexamethasone Intravitreal Implant for the Treatment of Macular Edema Following Retinal Vein Occlusion: Post Hoc Analysis of Post-Marketing Surveillance Data in the Real-World Setting in Korea. Clin Ophthalmol. 2021 Aug 27;15:3623-3636. doi: 10.2147/OPTH.S302014. eCollection 2021. PMID 34475750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Enrolled Population includes all 724 patients consented. The Safety Analysis Population includes 718 patients who were treated per protocol and completed a survey. The Safety Analysis Population was used for all analyses.
Period: Overall Study
Arm/Group | OZURDEX®
Started | 724
Completed | 718
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: The Enrolled Population includes all 724 patients consented. The Safety Analysis Population includes 718 patients who were treated per protocol and completed a survey. The Safety Analysis Population was used for all analyses.
Arm/Group | OZURDEX®
Number analyzed (Participants) | 718
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.18 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 424
  Male | 294

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events or Adverse Drug Reactions
Description: An Adverse Event is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. An Adverse Drug Reaction is a harmful and unintended reaction that is incurred during routine administration or use of the drug, whose causal relationship with the drug cannot be excluded.
Time Frame: 4 Years
Population: Safety Population: all patients who were treated per protocol and completed a survey
Measure: Number; unit: Patients
Arm/Group | OZURDEX®
Number analyzed (Participants) | 718
Patients
  Adverse Events | 55
  Adverse Drug Reactions | 50

2. Secondary Outcome: Percentage of Patients With 15 or More Letter Improvement in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved and was considered 'effective'. The percentage of patients with at least a 15 or more letter improvement in BCVA in the study eye are presented.
Time Frame: 4 Years
Population: Efficacy Population: all patients who were treated per protocol who had data available for analysis
Measure: Number; unit: Percentage of Participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 691
Percentage of Participants | 94.36

ADVERSE EVENTS:
Description: The Safety Analysis Population includes patients treated with dexamethasone 700 ㎍ (OZURDEX®) intravitreal implant and completed a survey. The Safety Analysis Population was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | OZURDEX®
Serious Adverse Events (participants affected / at risk) | 4/718
Other Adverse Events (participants affected / at risk) | 0/718
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=718)
Ocular Tension Decreased (Eye disorders) | 1
Endophthalmitis (Eye disorders) | 2
Macula Lutea (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.